CLINICAL TRIAL: NCT05924529
Title: ADRD Prevalence in American Samoa
Brief Title: Alzheimer's Disease and Related Dementias (ADRD) Prevalence in American Samoa
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: American Samoa Community Cancer Coalition (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Miami (Other); University of California, San Francisco (Other); University of Hawaii (Other)
Responsible Party: Sponsor
Other Study IDs: ASCCC0191792
Record Dates: First submitted 2023-02-27; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer's Disease and Related Dementia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will collect blood samples from participants in which some whole blood will be spun down for plasma extraction, some of it will be sent in whole blood form to a laboratory for analysis and the remaining will be stored in repository.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Samoans in American Samoa: Cognitive assessments will be administered to all participants to assess cognitive status. Gold standard evaluations will be administered to cross-validate the results of the cognitive assessments. Blood will be extracted from all participants to cross-validate results from the prior cognitive assessments and Gold Standard evaluations and conduct plasma and genetic analysis.

SUMMARY:
The goal of this study is to learn about ADRD prevalence within the Samoan population. Participants will be administered a series of cognitive assessments to determine cognitive status and a population-based prevalence of Mild Cognitive Impairment (MCI) and ADRD. Blood samples will also be collected from the participants for genetic and plasma biomarker analysis.

DETAILED DESCRIPTION:
This study aims to do the following:

Test ADRD knowledge, health literacy, research readiness and determine ADRD resilience and vulnerability factors, and cognitive status in a probability sample of 981 Samoans age 50+ using culturally adapted instruments in our probability sample.

Conduct Gold Standard evaluations in our probability sample using the Uniform Data Set (UDSv3.0) from the National Institute on Aging (NIA) Alzheimer's Disease Research Center program to determine a population-based prevalence of MCI and ADRD for harmonization, data sharing, and comparison to other groups, and,

Cross-validate Gold Standard dementia evaluations with genetic (i.e., ApoE) and plasma Amyloid-Tau-Neuronal Injury/Neurodegeneration (ATN) framework biomarkers in our probability sample and compare to information available for other racial/ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* Community dwelling
* Speaks English or Samoan
* Willing to contribute a biomarker specimen

Exclusion Criteria:

* Residing in Assistant Living or Skilled Nursing Facility
* Axis 1 Psychiatric diagnosis (e.g., Schizophrenia, Bipolar)
* Unstable medical condition (i.e., metastatic cancer) that could preclude completion of study visit

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: American Samoa is the only U.S. territory located south of the equator. The 2020 U.S. Census recorded 46,366 residents, with 11,025 (23.8%) of the population age 50 and over. Healthcare in American Samoa is extremely limited with only three government health care providers: 1 hospital, 5 Federally Qualified Health Centers, and Department of Human and Social Services providing WIC, mental health, and nutritional assistance programs. There are only a handful of private healthcare practices: 1 dentist, 2 primary care doctors, and 1 chiropractor. There are no neurologists in American Samoa and only 3 psychiatrists. There is no PET or MRI. There are no known studies documenting ADRD prevalence in the American Samoan population.
Sampling Method: Probability Sample
Enrollment: 1098 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Demographic Information and Socioeconomic Status | Demographic information collected will be assessed up to 1 year from when it was collected.
  Information on sociodemographic, primary language, medical and injury history, review of systems, medications, alcohol/tobacco/substance use history, exposure history, co-morbidities, social and family history are collected to determine the socioeconomic status of the participant. Socioeconomic status is determined by calculating the combined education and occupation attainment scores from the Hollingshead Two-Factor Index. This information will be aggregated to understand the socioeconomic status of the participant.
Charlson Comorbidity Index | Charlson co-morbidities will be assessed up to 1 year from when it was collected.
  The Charlson Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis codes. Each comorbidity category has an associated weight (from 1 to 6) and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
Functional Comorbidity Index (FCI) | Functional Comorbidities will be assessed up to 1 year from when it was collected.
  The Functional Comorbidity index (FCI) has been designed specifically in relation to physical function and is easier and more intuitive to use. It includes 18 diagnoses, counting their presence or absence, resulting in a cumulative sum score: the number of comorbidities.
Modified CAID System | mCAIDE index will be assessed up to 1 year from when it was collected.
  Modified CAIDE (mCAIDE) system and test its ability to predict presence, severity, and etiology of cognitive impairment in older adults. Higher mCAIDE quartiles were associated with lower performance on global and domain-specific cognitive tests.
ADRD Health Literacy | DeLA will be assessed up to 1 year from when it was collected.
  Dementia Literacy Assessment (DELA) consists of 25 items scored 0=incorrect/1=correct. Total DELA score ranges from 0 to 25 with a higher score being indicative of greater dementia literacy.
Quick Physical Activities Rating | QPAR score will be assessed up to 1 year from the date data was collected.
  The Quick Physical Activities Rating (QPAR) as an informant-rated instrument to quantify the dosage of physical activities in healthy controls. The higher the score, the better the participant's physical activity is. The lower the score, the lower the participant's physical activity.
MIND Diet | MIND Diet score will be assessed up to 1 year from the date data was collected.
  A MIND diet score was developed to identify foods and nutrients, along with daily serving sizes, related to protection against dementia and cognitive decline. The MIND diet identified fifteen dietary components that were classified as either "brain healthy" or as unhealthy. Participants with the highest MIND diet scores had a significantly slower rate of cognitive decline compared with those with the lowest scores.
Applied Mindfulness Process Scale | MIND Diet score will be assessed up to 1 year from the date data was collected.
  The Applied Mindfulness Process Scale (AMPS) is a process measure used to quantify how participants in mindfulness-based interventions (MBIs) use mindfulness practice when facing challenges in daily life.
ADRD Vulnerability | The VI scores will be assessed up to 1 year from the date the data was collected.
  The Vulnerability Index (VI) was designed to identify individuals who are at risk of developing cognitive impairment in the future, capturing 12 sociodemographic variables and modifiable medical comorbidities associated with higher ADRD risk.
  A weighted measure of the contributions of age, sex, race, education, depression, blood pressure, obesity, diabetes, stroke, heart disease, hypercholesterolemia, and frailty to ADRD risk.
  The VI has the possible range of scores from 2-20 with higher scores representing higher brain vulnerability with a published cut-off of 8.
Quick Dementia Rating Scale | Quick Dementia Rating Scale score will be assessed up to 1 year from the date the data was collected.
  The Quick Dementia Rating Scale is a 10-item questionnaire completed by an informant without the need for a trained clinician or rater, and takes 3 to 5 minutes to complete. Scores range from 0 to 30 with higher scores representing greater cognitive impairment.
Number Symbol Coding Task | Number Symbol Coding Task score will be assessed up to 1 year from the date the data was collected.
  The Number Symbol Coding Task is a brief, 90-second executive task that incorporates attention, planning and set-switching that can be completed by individuals into the moderate-to-severe stages of dementia.
  The Number Symbol Coding Task score are between 0-70 where higher scores can distinguish between normal controls, MCI and ADRD.
Dementia Screening Platform | Scores that constitute the dementia screening platformed will be assessed up to 1 year from the date the data was collected.
  The platform combines the QDRS, NSCT, RI and VI to discriminate between normal controls, MCI and ADRD.
Montreal Cognitive Assessment (MoCA) | Scores of the MoCA-B will be assessed 1 year from the date the data was collected.
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible score is 30 points; a score of 26 or above is considered normal.
Cognivue Clarity | Cognivue clarity scoare will be assessed 1 year from the date the data was collected.
  Cognivue Clarity evaluates 6 cognitive domains: visuospatial, executive function/attention, naming/language, memory, delayed recall and abstraction. Cognivue Clarity also measures two speed performance parameters: reaction time and speed processing. Scores that ≥ 75: Normal Cognitive Function, 51-74: Low Cognitive Impairment and ≤ 50: Moderate-Severe Cognitive Impairment.
Demographic Information | Demographic information of the participant will be taken 90 days from the day they took the MoCA administered initially.
  Updated information on sociodemographic data using UDSv3.0 forms.
Medical Evaluation | Medical evaluation should be completed within 90 days from the day the MoCA was administered.
  A physical and neurological examination will be completed in which the Modified Hachinski Scale will be used to assess vascular risks. Participants scoring 7 or greater are classified as having "multi-infarct dementia", and patients scoring </= 4 are classified as having "primary degenerative dementia". A score of 5 or 6 is considered as an intermediate value and is usually designated as "mixed dementia".
MINT Evaluation | MINT score should be completed and assessed within 90 days from the day the MoCA was administered.
  The Multilingual Naming Test (MINT) is a picture naming test to detect naming impairment (i.e., dysnomia) across stages of Alzheimer's disease (AD). The number of spontaneous correct responses and correct responses following a semantic cue are summed to give a total score. Thus, the abbreviated MINT total scores range from 0 to 32 and these were used as the primary outcome measure.
  Individuals with a low score on MINT are generally less effective and tend to exhibit undesirable behaviors such as unauthorized absence, inappropriate behavior and an irresponsible approach to rules and regulations.
  People with a high score at MINT are generally considered to be high-performing, both in the handling of work tasks and working relationships.
Craft Story Evaluation | Cognitive evaluation should be completed within 90 days from the day the MoCA was administered.
  Craft story immediate, delayed and cued paragraph recall assesses the ability to recall a short story that was read to them 20 minutes ago.
Benson Copy Evaluation | Cognitive evaluation should be completed within 90 days from the day the MoCA was administered.
  Benson Copy assesses visuospatial and constructional ability/skills. Benson Copy Test
Category and Letter fluency Evaluation | Cognitive evaluation should be completed within 90 days from the day the MoCA was administered.
  Category and Letter fluency assesses verbal fluency and language (semantic memory).
Number Forward/Backward Evaluation | Cognitive evaluation should be completed within 90 days from the day the MoCA was administered.
  Number forward measures capacity for holding information briefly for the purpose of repeating exactly.
  Number backward measures ability to hold information and manipulate the numbers by reversing the sequence.
Trailmaking A & B Evaluation | Cognitive evaluation should be completed within 90 days from the day the MoCA was administered.
  Trailmaking A & B assesses attention/processing speed, and executive function/cognitive flexibility.
  Activity:
  Part A - The examiner instructs the participant to connect the circles (number 1 through 25) with a drawn line in ascending order as quickly as possible.
  Part B - The examiner instructs the participant to connect alphanumeric circles with a drawn line in ascending order as quickly as possible.
Noise Pareidoloia Evaluation | Cognitive evaluation should be completed within 90 days from the day the MoCA was administered.
  Noise-Pareidoloia Test is a tool that evokes visual hallucination-like illusions, and these illusions may be a surrogate marker of visual hallucinations.
Geriatric Depression Evaluation | Cognitive evaluation should be completed within 90 days from the day the MoCA was administered.
  Geriatric Depression Scale is a patient-reported outcome measure created to screen for depressive symptoms among older adults. The GDS is a multidimensional, multidisciplinary diagnostic and therapeutic activity that helps find patients at risk of/with depression.
  Scores of 1 to 5 is normal. Higher scores suggests more depression.
Functional Activities Questionnaire | Cognitive evaluation should be completed within 90 days from the day the MoCA was administered.
  Functional Activities Questionnaire to assess activities of daily living.
Neuropsychiatric Inventory | Cognitive evaluation should be completed within 90 days from the day the MoCA was administered.
  Neropsychiatric Inventory to assess behavior.
Plasma Amyloid-β42 | Plasma evaluation should be completed within 90 days from the day the MoCA was administered.
  ADRD plasma biomarkers will be analyzed by MagQu Ltd to measure plasma Aβ42 using the Simoa Human assays (Quanterix Corporation, Billerica, MA) on the Simoa™ HD-X. The 42 amino acid form of amyloid-β (Aβ42) plays a key role in the pathogenesis of Alzheimer's disease (AD) and is a core biomarker for the diagnosis of AD.
Plasma Amyloid-β40 | Plasma evaluation should be completed within 90 days from the day the MoCA was administered.
  ADRD plasma biomarkers will be analyzed by MagQu Ltd to measure plasma Aβ40 using the Simoa Human assays (Quanterix Corporation, Billerica, MA) on the Simoa™ HD-X. Amyloid β (Aβ) is known as a biomarker for AD, and the CSF Aβ40 / Aβ42 ratio is clinically useful for diagnosis of AD.
Plasma P-tau181 | Plasma evaluation should be completed within 90 days from the day the MoCA was administered.
  ADRD plasma biomarkers will be analyzed by MagQu Ltd to measure p-tau-181 using the Simoa Human assays (Quanterix Corporation, Billerica, MA) on the Simoa™ HD-X to measure neuronal injury. Plasma P-tau181 is a noninvasive diagnostic and prognostic biomarker of AD.
Glial Fibrillary Acidic Protein | Plasma evaluation should be completed within 90 days from the day the MoCA was administered.
  ADRD plasma biomarkers will be analyzed by MagQu Ltd to measure Glial Fibrillary Acidic Protein using the Simoa Human assays (Quanterix Corporation, Billerica, MA) on the Simoa™ HD-X to measure neuronal injury.
Neurofilament Light | Plasma evaluation should be completed within 90 days from the day the MoCA was administered.
  ADRD plasma biomarkers will be analyzed by MagQu Ltd will measure neuronal injury neurofilament light with the Simoa Human assays (Quanterix Corporation, Billerica, MA) on the Simoa™ HD-X.
Synuclein | Plasma evaluation should be completed within 90 days from the day the MoCA was administered.
  ADRD plasma biomarkers will be analyzed by MagQu Ltd will measure Alpha Synuclein using the Simoa™Human assays (Quanterix Corporation, Billerica, MA) on the Simoa™ HD-X.
Genetics | Genetic evaluation should be completed within 90 days from the day the MoCA was administered.
  We will conduct several analyses taking in account the limitations of small sample size, including genotyping, whole genome sequencings (WGS), preliminary novel gene variant exploration, and local ancestry. All samples will be genotyped using GSA Illumina array at the HIHG Center for Genome Technology (CGT)

CONTACTS AND LOCATIONS:
Overall Officials: Va'atausili Tofaeono, MS, Principal Investigator — American Samoa Community Cancer Coalition
Locations (2):
- American Samoa (2):
  - Malaloa GHC Reid Building, Pago Pago
  - Sa'o Fetalai Building, Pago Pago

IPD SHARING:
Plan to Share IPD: Yes
The Multi Principal Investigators are committed to placing its data in the public domain where it will be available to qualified scientific investigators by a defined process and at time intervals, in accordance with NIH policy. The database/registry may be very attractive for the evaluation of potential therapies for age-related diseases. the database will: 1) serve pedagogy (education) functions, 2) facilitate standardized collection and analysis protocols, and 3) promote collaboration among investigators (within and between institutions). We have a web-based resource repository developed and an account at Open Science Framework and upon acceptance of a publication, a de-identified dataset (including any genetic data) with all variables related to that publication will be placed at Open Science Framework and a Digital Object Identifier will be made available in all publications following HIPAA and Institutional Review Board guidelines.
Supporting Information: CSR
Time Frame: After study has been completed.
Access Criteria: The database may be attractive for the evaluation of prevalence, impact, and potential therapies for age-related diseases. We will develop a process wherein formal proposals to conduct clinical trials or other studies with the cohort are evaluated and approved.

REFERENCES:
- [Background] Tofaeono V, Ka'opua LSI, Sy A, Terada T, Taliloa-Vai Purcell R, Aoelua-Fanene S, Tong K, Tofaeono V, Unutoa-Mageo T, Scanlan L, Cassel K, Rosario A. Research Capacity Strengthening in American Samoa: Fa'avaeina le Fa'atelega o le Tomai Sa'ili'ili i Amerika Samoa. Br J Soc Work. 2020 Mar;50(2):525-547. doi: 10.1093/bjsw/bcz160. Epub 2019 Dec 31. PMID 32280149
- [Background] Williams S, Graupner J, Fernandes R, Gorawara-Bhat R. Healthcare providers attitudes and knowledge toward dementia in American Samoan culture. J Pain Sym Man 55:P680, 2017

DOCUMENTS (1):
  • Informed Consent Form (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT05924529/ICF_000.pdf